CLINICAL TRIAL: NCT02074566
Title: A Prospective Randomized Multicentre Efficacy Study on Defining the Optimal Cryoballoon Duration Therapy for Treatment of Atrial Fibrillation: The 1-2-3 Study
Brief Title: Defining the Optimal Cryoballoon Duration Therapy for Treatment of Atrial Fibrillation: Defining the Optimal Cryoballoon Duration Therapy for Treatment of Atrial Fibrillation: The 1-2-3 Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Harald Verheij (Other)
Collaborators: Thorax Centrum Twente (Other); Academisch Ziekenhuis Maastricht (Other)
Responsible Party: Sponsor-Investigator, Harald Verheij, Drs., Thorax Centrum Twente
Organization: Thorax Centrum Twente (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: NL47337.044.13
Record Dates: First submitted 2014-02-10; First posted 2014-02-28 (Estimated); Last update posted 2020-03-12 (Actual); Status verified 2019-04

CONDITIONS: Atrial Fibrillation
Keywords: Pulmonary Vein Isolation; Atrial fibrillation; Cryoballoon therapy; Duration
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (3):
- 2 times 1 (Other): PVI will be performed using a cryoballoon ablation application time of 2 times 1 minute
  Interventions: Other: Cryoballoon ablation
- 2 times 2 (Other): PVI will be performed using a cryoballoon ablation application time of 2 times 2 minutes
  Interventions: Other: Cryoballoon ablation
- 2 times 3 (Other): PVI will be performed using a cryoballoon ablation application time of 2 times 3 minutes
  Interventions: Other: Cryoballoon ablation

INTERVENTIONS:
Other: Cryoballoon ablation — PVI using cryoballoon

SUMMARY:
Cryoballoon based therapy is an established therapy for the treatment of (paroxysmal) atrial fibrillation. However, with the rapid evolution in cryoablation technique and its increased effectiveness, the risk of complications increases. Therefore it is of utmost importance to define the optimal duration of cryoballoon ablation time.The objective of the study is to assess the optimal ablation duration using the second generation cryoballoon for isolation of pulmonary veins in the treatment of atrial fibrillation.

DETAILED DESCRIPTION:
Rationale Cryoballoon based therapy is an established therapy for the treatment of (paroxysmal) atrial fibrillation. However, with the rapid evolution in cryoablation technique and its increased effectiveness, the risk of complications increases. Therefore it is of utmost importance to define the optimal duration of cryoballoon ablation time.

Objective To assess the optimal ablation duration using the second generation cryoballoon for isolation of pulmonary veins in the treatment of atrial fibrillation.

Study design The study is designed as a prospective multicentre randomized efficacy study.

Study population Patients 18-70 years of age with paroxysmal atrial fibrillation eligible for pulmonary vein isolation according to current international guidelines.

Intervention Patients will be randomized to 2 cycles of 1, 2 or 3 minutes of cryoballoon ablation after reaching the temperature "plateau phase".

Main study parameters/endpoints Acute success of pulmonary vein isolation.

Nature and extent of the burden and risks associated with participation, benefit and group relatedness:

No additional risk is present as the procedure is common clinical practice, current cryoballoon application time is 3 minutes Shorter application times are not expected to add to the risk.

ELIGIBILITY:
Inclusion Criteria:

* Paroxysmal atrial fibrillation eligible for pulmonary vein isolation according to current international guidelines.
* Age < 70 years.
* Willing and able to sign informed consent.
* Willing to and capable of following the requested study procedures.

Exclusion Criteria:

* Age < 18 years.
* Pregnancy
* Life or follow-up expectancy < 12 months.
* Previous PVI.
* Contrast allergy.
* Creatin clearance level < 60.
* Left ventricular ejection fraction < 40%
* Abnormal left atrium anatomy defined as number of PV's ≠ 4 or Left Atrium diameter >50mm (measured in the parasternal long axis, as assessed with transthoracic echocardiography) or >40 cc/m2 . This will lead to exclusion after inclusion but before randomisation.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 222 (Actual)
Dates: Start 2014-08-14 (Actual); Primary Completion 2018-03-08 (Actual); Study Completion 2019-02-13 (Actual)

PRIMARY OUTCOMES:
Number of patients wit successfull pulmonary vein isolation | up to 6 minutes
  Assessment of successfull pulmonary vein isolation after 2 x 1/2/3 minutes of cryoballoon application. The assessment of this outcome will take place during the procedure.

SECONDARY OUTCOMES:
Number of complications | 1 year
  Complications being:
  1. Phrenic nerve palsy or diminishment of diaphragm excursion during cryo-ablation.
  2. Temperatures reaching <12 C in the oesophagus during cryoablation.
  3. Other complications such as delayed gastric emptying, pericardial fluid/tamponade, haemoptoe, vascular complications.
Patients in which acute success of pulmonary vein isolation (after 1 freezing cycle) was present | up to 6 minutes
  The assessment of this outcome will take place during the procedure
Duration of thaw phase (= time between end of freezing to automatic deflation of the balloon) related to acute success of pulmonary vein isolation | up to 6 minutes
  The assessment of this outcome will take place during the procedure.
Procedure time, fluoroscopy time, amount of contrast used | up to 6 minutes
  The assessment of this outcome will take place right after the procedure. It measures procedural parameters.
Lower Esophageal Temperature development | up to 6 minutes
  The measurement will take place during the procedure. It registrates the lower esophageal temperature ande the development during the course of the procedure.
Atrial Fibrillation recurrence | after 1 year follow up
Balloon temperatures measured by the console | up to 6 minutes

CONTACTS AND LOCATIONS:
Locations (2):
- Netherlands (2):
  - Medisch Spectrum Twente, Enschede, Nederland
  - Maastricht University Medical Centre, Maastricht